CLINICAL TRIAL: NCT03064035
Title: A Prospective, Randomized Study of Fixed Versus Variable Dosing of 4-factor Prothrombin Complex Concentrate for Emergent Warfarin Reversal at a Large Tertiary Care Medical Center
Brief Title: Fixed Versus Variable Dosing of 4-factor Prothrombin Complex Concentrate for Emergent Warfarin Reversal
Acronym: kcentra
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A16-732
Record Dates: First submitted 2017-02-16; First posted 2017-02-24 (Actual); Results first posted 2023-07-11 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2019-06

CONDITIONS: Acute Bleeding on Long-Term Anticoagulation Therapy; Hemorrhage; Significant Bleeding in Patients With a Coagulopathy (Prolonged Thrombin Time); Urgent Reversal of Vitamin K Antagonist (VKA) Anticoagulation
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Intervention Model Description: For adults on long-term warfarin therapy who present to the ED with emergent bleeding, or who are in need of urgent invasive surgical procedures: the exposure of interest will be fixed vs. variable dose 4FPCC, to which eligible patients will be randomly assigned in a 1:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fixed dose 4FPCC (Experimental): Incorporating a fixed dose of 1500 IU.
  If the patient receiving the 1500 IU fixed dose remains in a bleeding state and the INR remains above goal, an additional 500 IU may be administered at the physician's discretion to minimize bleeding and attempt to achieve hemostasis.
  Interventions: Drug: 4-factor prothrombin complex concentrate (4FPCC)
- Variable dose 4FPCC (Active Comparator): The FDA-approved variable dosing algorithm is as follows:
  initial INR 2-3.9: 25 IU/kg (maximum dose 2500 IU), initial INR 4-6: 35 IU/kg (maximum dose 3500 IU), and initial INR >6: 50 IU/kg (maximum dose 5000 IU). The patient weight will be obtained using a scale and documented by the treating registered nurse
  Interventions: Drug: 4-factor prothrombin complex concentrate (4FPCC)

INTERVENTIONS:
Drug: 4-factor prothrombin complex concentrate (4FPCC) — 4-factor prothrombin complex concentrate (4FPCC) contains all of the vitamin K-dependent clotting factors inhibited by warfarin, making it desirable for use in warfarin reversal for emergent bleeds. Multiple guidelines currently recommend 4FPCC for warfarin reversal in vitamin K-dependent major bleeding or intracranial hemorrhage. 4FPCC has a fast onset of action and has demonstrated significant reversal of INR within 10 minutes. Its duration of action is up to 8 hours, and for this reason it should be given concurrently with vitamin K. Vitamin K has a delayed onset of action due to its need to stimulate the synthesis of clotting factors so its effects begin as the effects of 4FPCC diminish. 4FPCC is the standard of care treatment for this clinical population in the Regions Hospital Emergency Department.

SUMMARY:
The goal of this study is to determine if a fixed dose of 4-factor prothrombin complex concentrate (4FPCC) is as effective as the current standard of care. 4FPCC is used to reverse the effects of warfarin when a patient has emergent bleeding. The investigators hope that this study will help doctors treat patients quicker in the future. In addition, it may be cheaper for patients and hospitals. This is the same medication the doctor would use to reverse warfarin's effects, but at a lower dose.

Hypothesis: A fixed dose of 4FPCC will be comparable to FDA-approved variable dosing for reversal of warfarin-induced anticoagulation (defined as an international normalized ratio [INR] ≤ 1.5) in patients with an INR ≥2 experiencing an emergent bleed or requiring emergent surgery.

DETAILED DESCRIPTION:
Warfarin is a common oral anticoagulant utilized in the United States for the treatment and prevention of thromboembolic events and conditions. Although effective, the major complication associated with warfarin is the risk of major bleeding events. Incidence of major bleeding events in long-term warfarin users is 1.5% to 5.2% per year, with mortality exceeding 13%. Among patients with an intracranial bleed, the mortality rate increases to 46%-55%. In these situations, it is imperative to reverse the pharmacologic effects of warfarin quickly in order to minimize bleeding and reduce the risk of death. Warfarin inhibits formation of vitamin K-dependent clotting factors II, VII, IX, X, and proteins C and S. An international normalized ratio (INR) is a commonly utilized laboratory test to measure the amount of anticoagulation provided by warfarin and is monitored throughout therapy. The INR is a standardized ratio utilizing prothrombin time to prevent variation between institutional laboratories. Prothrombin time is defined as the time required for plasma to clot after addition of clotting factor. A normal INR in a healthy adult can range from 0.8-1.2. The majority of patients on chronic warfarin therapy will have a target INR of 2-3.

The optimal dose of 4FPCC is currently unknown despite multiple studies evaluating different dosing regimens. The FDA-approved dosing is 25 to 50 IU factor IX per kilogram of body weight, depending on INR. It is dosed to a maximum of 100 kilograms of body weight. The FDA-approved variable dosing algorithm is as follows: initial INR 2-3.9: 25 IU/kg (maximum dose 2500 IU), initial INR 4-6: 35 IU/kg (maximum dose 3500 IU), and initial INR >6: 50 IU/kg (maximum dose 5000 IU). Exact doses of 4FPCC administered may vary slightly from the calculated doses as the amount of 4FPCC differs based on the vials utilized.

By incorporating a fixed dose of 1500 IU, presenting INR and body weight may not need to be determined prior to administration. This may allow for early administration and prevent delay for warfarin reversal in patients with emergent bleeding. This research may determine whether a fixed dose is effective for reversing warfarin to a target INR less than 1.5 compared to FDA-approved variable dosing. In addition, the lower fixed-dose will significantly reduce costs to the institution.

Hypothesis: A fixed dose of 4FPCC will be comparable to FDA-approved variable dosing for reversal of warfarin-induced anticoagulation (defined as an international normalized ratio [INR] ≤ 1.5) in patients with an INR ≥2 experiencing an emergent bleed or requiring emergent surgery.

ELIGIBILITY:
Inclusion Criteria:

* Chronic anticoagulation with warfarin and initial INR ≥2
* Emergent bleeding (i.e. intracranial hemorrhage, gastrointestinal hemorrhage, urgent invasive procedures, etc.) or urgent surgery requiring reversal of INR to ≤1.5

Exclusion Criteria:

* Younger than 18 years of age
* History of heparin-induced thrombocytopenia (HIT)
* Patients without initial or post-administration INR readings
* Patients with an initial INR <2
* Pregnant patients
* Prisoners

Ages: 18 Years to 125 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Stoecker, PharmD, Principal Investigator — Regions Hospital
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total 192 patients who presented to the emergency department with emergent bleeding were screened for eligibility and 79 of these patients were enrolled. 107 did not meet inclusion criteria, 1 declined participation, and 5 were unable to be enrolled prior to administration of Kcentra.
Groups:
- Fixed Dose 4FPCC: Incorporating a fixed dose of 1500 IU.
  If the patient receiving the 1500 IU fixed dose remains in a bleeding state and the INR remains above goal, an additional 500 IU may be administered at the physician's discretion to minimize bleeding and attempt to achieve hemostasis.
  4-factor prothrombin complex concentrate (4FPCC): 4-factor prothrombin complex concentrate (4FPCC) contains all of the vitamin K-dependent clotting factors inhibited by warfarin, making it desirable for use in warfarin reversal for emergent bleeds. Multiple guidelines currently recommend 4FPCC for warfarin reversal in vitamin K-dependent major bleeding or intracranial hemorrhage. 4FPCC has a fast onset of action and has demonstrated significant reversal of INR within 10 minutes. Its duration of action is up to 8 hours, and for this reason it should be given concurrently with vitamin K. Vitamin K has a delayed onset of action due to its need to stimulate the synthesis of clotting factors so its effects begin as the effects of 4FPCC diminish. 4FPCC is the standard of care treatment for this clinical population in the Regions Hospital Emergency Department.
- Variable Dose 4FPCC: The FDA-approved variable dosing algorithm is as follows:
  initial INR 2-3.9: 25 IU/kg (maximum dose 2500 IU), initial INR 4-6: 35 IU/kg (maximum dose 3500 IU), and initial INR >6: 50 IU/kg (maximum dose 5000 IU). The patient weight will be obtained using a scale and documented by the treating registered nurse
  4-factor prothrombin complex concentrate (4FPCC): 4-factor prothrombin complex concentrate (4FPCC) contains all of the vitamin K-dependent clotting factors inhibited by warfarin, making it desirable for use in warfarin reversal for emergent bleeds. Multiple guidelines currently recommend 4FPCC for warfarin reversal in vitamin K-dependent major bleeding or intracranial hemorrhage. 4FPCC has a fast onset of action and has demonstrated significant reversal of INR within 10 minutes. Its duration of action is up to 8 hours, and for this reason it should be given concurrently with vitamin K. Vitamin K has a delayed onset of action due to its need to stimulate the synthesis of clotting factors so its effects begin as the effects of 4FPCC diminish. 4FPCC is the standard of care treatment for this clinical population in the Regions Hospital Emergency Department.
Period: Overall Study
Arm/Group | Fixed Dose 4FPCC | Variable Dose 4FPCC
Started | 39 (Randomized to fixed dosing) | 40 (Randomized to variable dosing)
Completed | 34 (Fixed dosing subjects used in analysis) | 37 (Variable dosing subjects used in analysis)
Not Completed | 5 | 3
Not completed — Did not receive allocated intervention | 4 | 2
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Patients were randomized to one of two arms - fixed or variable dosing
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed Dose 4FPCC | Variable Dose 4FPCC | Total
Number analyzed (Participants) | 34 | 37 | 71
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: There are two different age ranges based on randomized groups - fixed and variable dosing
  years | 74.5 [62.5 to 86.5] | 76 [67.5 to 84.5] | 76 [65.5 to 86.5]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There are two different sex distributions for the two randomized groups - fixed and variable dosing
  Participants
    Female | 10 | 13 | 23
    Male | 24 | 24 | 48
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: There are two different randomized groups - fixed and variable dosing
  participants
    United States | 34 | 37 | 71

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Demonstrated Significant Reversal of INR Within 15 Minutes
Description: To evaluate whether fixed dose 4FPCC is acceptably comparable to variable dosing with respect to anticoagulation reversal, as defined by a targeted INR of ≤1.5
Time Frame: 15 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Dose 4FPCC | Variable Dose 4FPCC
Number analyzed (Participants) | 34 | 37
Participants | 21 | 33

2. Secondary Outcome: Number of Participants With a Thromboembolic Event
Description: Study patients will be followed post-administration of 4FPCC for thromboembolic events such as deep vein thrombosis, pulmonary embolism, ischemic stroke or transient ischemic event, or myocardial infarction.
Time Frame: up to 7 days post administration of 4FPCC
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Dose 4FPCC | Variable Dose 4FPCC
Number analyzed (Participants) | 34 | 37
Participants | 0 | 0

3. Secondary Outcome: Total Cost of Dosing Strategy
Description: Cost outcomes will be assessed for all study patients and compared by dosing assignment. Cost of treatment was assessed based on the amount of 4FPCC doses administered during admission, using the study-contemporary rate of $1.57/unit
Time Frame: Hospital Stay, Up to 6 months
Measure: Median (Inter-Quartile Range); unit: dollars
Arm/Group | Fixed Dose 4FPCC | Variable Dose 4FPCC
Number analyzed (Participants) | 34 | 37
dollars | 2524.56 [2497.87 to 2551.25] | 3372.36 [2643.36 to 4101.36]

ADVERSE EVENTS:
Time Frame: From enrollment through 7 days.
Arm/Group | Fixed Dose 4FPCC | Variable Dose 4FPCC
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/37
Other Adverse Events (participants affected / at risk) | 0/34 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT03064035/Prot_SAP_001.pdf